CLINICAL TRIAL: NCT01030887
Title: Individually Prescribed Exercise Versus Usual Care in a Heterogeneous Cancer Survivor Population: A Pragmatic Randomized Controlled Trial
Brief Title: PEACH Trial: Prescribed Exercise After Chemotherapy
Acronym: PEACH
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Dublin, Trinity College (Other)
Collaborators: Health Research Board, Ireland (Other)
Responsible Party: Julie Walsh, Trinity College Dublin
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CTPF/2008/12
Record Dates: First submitted 2009-12-11; First posted 2009-12-14 (Estimated); Last update posted 2011-08-15 (Estimated); Status verified 2009-11

CONDITIONS: Cancer
Keywords: Cancer; Exercise; Physical Activity; Randomized controlled trial
MeSH Terms: conditions — Neoplasms; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Exercise Programme (Active Comparator): This will consist of an 8-week exercise programme, performed twice per week.
  Interventions: Behavioral: Exercise programme
- Usual Care (Placebo Comparator): Standard practice including opportunistic exercise advice and patients' self-directed physical activity
  Interventions: Behavioral: Exercise programme

INTERVENTIONS:
Behavioral: Exercise programme — Moderate intensity exercise

SUMMARY:
Many cancer survivors suffer symptoms such as fatigue and dyspnea which may persist for years or months after their chemotherapy has finished. Despite the known benefits of exercise and its potential to address many of the symptoms after cancer, the type of practical exercise programme which best suits this population is not known.

Many exercise programmes performed in cancer survivors take place over many weeks or months and include people with specific types of cancer. Such programmes may therefore not be suitable for the majority of cancer survivors and would pose serious practical difficulties with high drop-out rates and expensive resource consumption if they were extended into clinical practice.

We propose to run an 8-week exercise intervention in a mixed cancer population.

Hypothesis: A brief, individually tailored 8-week intervention will increase fitness and improve other physical symptoms in a mixed cancer survivor population after chemotherapy.

DETAILED DESCRIPTION:
Background: Many cancer survivors suffer a range of physical and psychological symptoms with may persist for years or months after treatment finishes. Despite the known benefits of exercise and its potential to address many of these adverse effects of treatment, the role of exercise as well as its optimum duration, frequency, and intensity in this population has yet to be fully elucidated. Many cancer rehabilitation programmes presented in the literature are very long, have tight eligibility criteria and are not likely to be practical in the majority of cancer survivors. We plan to investigate a novel brief 8-week intervention which aims to increase physical fitness, and address other physical symptoms in a heterogeneous cancer survivor population.

Methods/design: Approximately 60 cancer survivors 2-6 months after completion of chemotherapy, usually adjuvant, with curative intent will be recruited through oncology clinics in a single institution and randomised to usual care or an exercise intervention. The exercise intervention consists of two specifically tailored, supervised, moderate intensity aerobic exercise sessions per week for 8 weeks. All participants will be assessed at baseline (0 weeks), post intervention (8 weeks), and at 3-month follow-up. The primary outcome measure is fitness, and secondary patient-related outcome measures include fatigue, quality of life, and morphological outcomes. A further secondary outcome is process evaluation including adherence to and compliance with the exercise program.

Discussion: This study will provide valuable information about the physical outcomes of this 8-week supervised aerobic programme. Additional process information and economic evaluation will inform the feasibility of implementing this program in a heterogeneous population after chemotherapy treatment with curative intent.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of solid tumour and completion of adjuvant chemotherapy (and/or radiotherapy) with curative intent within the preceding 2-6 months. (Patients who have received neoadjuvant chemotherapy or chemoradiotherapy followed by surgery will also be eligible. In addition, patients continuing onto adjuvant hormone therapy and anti-Her2 directed therapy are eligible).
* Ability to understand English
* Willing to be randomised
* Medical clearance to exercise
* Age 21-69
* Fitness level average, fair or poor according to certain pre-determined cut-off points for age and gender(Fletcher et al., 2001)
* Willing and able to attend supervised exercise sessions twice weekly for a period of 8 weeks, with an intention of achieving > 90% attendance
* LVEF > 50% and not < 20% worse than baseline in applicable patients

Exclusion Criteria:

* Evidence of active cancer
* Chronic medical and orthopaedic conditions that would preclude exercise (eg uncontrolled congestive heart failure or angina, recent MI, breathing difficulties requiring oxygen use or hospitalization)
* On beta-blocker medication
* Prior history of another cancer in previous 5 years (exception: non-melanoma skin cancer and non-invasive cancer of the cervix)
* Confirmed pregnancy
* Dementia or psychiatric illness that would preclude ability to participate in study
* Incomplete haematological recovery after chemotherapy (WCC< 3, Hb < 10 or Platelets < 100)
* BMI > 35
* LVEF post chemotherapy < 50% or > 20% deterioration of baseline pre-systemic treatment. LVEF criteria are applicable in patients who have received chemotherapy deemed in normal clinical practice to have a potential effect LVEF and in whom the LVEF will have been measured before systemic treatment and at end of chemotherapy

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2010-01; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Modified Bruce Treadmill Test (Fitness) | 0, 8 weeks, 3 months

SECONDARY OUTCOMES:
FACT-G scale (Quality of life-overall) | 0, 8 weeks, 3 months
FACT-F (Fatigue) | 0, 8 weeks, 3 months
RT3 Accelerometry (Activity level) | 0, 8 weeks, 3 months
Tanita Body Fat Assessment (% fat) | 0, 8 weeks, 3 months
SF-36v2 (Quality of life-functional aspects) | 0, 8 weeks and 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Dearbhaile O' Donnell, MD, Principal Investigator — St. James's Hospital, Dublin, Ireland; Juliette Hussey, PhD, Principal Investigator — Trinity College Dublin, Ireland; Julie M Walsh, MSc, Principal Investigator — University of Dublin, Trinity College
Locations (1):
- Medical Oncology Department, St. James's Hospital, Dublin, Ireland

REFERENCES:
- [Background] Walsh JM, Hussey J, Guinan E, O' Donnell D. 'Pragmatic randomized controlled trial of individually prescribed exercise versus usual care in a heterogeneous cancer survivor population': a feasibility study PEACH trial: prescribed exercise after chemotherapy. BMC Cancer. 2010 Feb 15;10:42. doi: 10.1186/1471-2407-10-42. PMID 20156345
- See also: Sponsor's web page — http://www.hrb.ie/
- See also: University affiliated to this research — http://www.tcd.ie/
- See also: Hospital affiliated to this research — http://www.stjames.ie/